CLINICAL TRIAL: NCT03853655
Title: Adjuvant Radiotherapy in Early Stage Oral Cancers (AREST)
Brief Title: Adjuvant Radiotherapy in Early Stage Oral Cancers
Acronym: AREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: NATIONAL CANCER GRID (Unknown)
Responsible Party: Principal Investigator, Dr. Sudhir Nair, Professor, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1713
Record Dates: First submitted 2017-06-20; First posted 2019-02-25 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cancer of Mouth; Cancer of the Tongue; Cancer of the Head and Neck; Buccal Mucosa Cancer; Floor of Mouth Carcinoma
Keywords: Cancer of the Mouth; Tongue cancer; Buccal Mucosa cancer; Head and Neck; Oral Cancer; Adjuvant Radiotherapy; Depth of Invasion
MeSH Terms: conditions — Mouth Neoplasms; Tongue Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (No Intervention): Patients in this arm will be observed and kept under active follow-up after surgery for the primary.
- Study arm (Experimental): Intervention in the study arm will be in the form of post-operative adjuvant radiotherapy starting within 6-weeks after primary surgery.
  Interventions: Radiation: Post-operative adjuvant radiotherapy

INTERVENTIONS:
Radiation: Post-operative adjuvant radiotherapy — Conventional treatment planning, as well as intensity-modulated radiation therapy (IMRT) planning, would be allowed on the study with patients being stratified on the RT technique.
  Treatment would be delivered on telecobalt unit (gamma-rays/linear accelerator (6MV photons). All fields would be treated daily.
  Phase I: 46 Gray(Gy) in 23 fractions over 4.5 weeks Phase II: 14Gray in 7 fractions over 1.5 weeks
  For IMRT, inverse planning would be done on a commercial TPS configured to deliver IMRT using 6MV photons. Patients shall be treated using the simultaneous integrated boost (SIB) technique with 5 fractions being delivered every week.
  Arms: Study arm

SUMMARY:
This study will assess the benefit of postoperative adjuvant radiotherapy in patients with an early oral squamous cell carcinoma (OSCC) having tumor thickness more than or equal to 5mm. The study population will consist of patients who have been treated by surgery for early stage oral tongue cancers. Patients with a close or positive margin (</= 5mm) and or with metastatic neck node(s) will be excluded. Selected patients will be randomized into two groups. The group I will be observed after surgery and group II will receive adjuvant radiotherapy as per protocol.

DETAILED DESCRIPTION:
The aim of this study is to assess the benefit of postoperative adjuvant radiotherapy in patients with an early oral squamous cell carcinoma (OSCC) having a tumor depth of invasion more than or equal to 5mm.

Primary objective:

To determine the impact of postoperative adjuvant radiotherapy on locoregional recurrence-free survival in patients with early-stage oral tongue cancer with tumor thickness ≥ 5 mm.

Secondary objectives:

1. To compare disease-free survival and overall survival between the two groups.
2. To assess and compare the quality of life changes between the two groups.
3. To assess the acute and long-term radiation toxicity.

We will be conducting a Phase III Open-Label Prospective Randomized Controlled Trial using stratified randomization. Patients will be randomized into two groups:

Group I: Control arm (Observation only) Group II: Study arm (Postoperative adjuvant radiotherapy)

Patients will be stratified on the following factors

1. Presence of Perineural Invasion (PNI)/Lympho-Vascular Emboli (LVE)
2. Histological grade (well-differentiated/moderately differentiated vs poorly differentiated)
3. Tongue/Floor of Mouth vs Buccal Mucosa.

Study procedures:

The study population will consist of patients who have been treated by surgery for early-stage oral cancers. Patients satisfying the inclusion-exclusion criteria will be included in the study after obtaining a valid, written and informed consent. The depth of invasion will be assessed microscopically by measuring the maximum vertical bulk of the tumor from the normal mucosal surface to the deepest point of invasion. After reviewing the histopathological report, patients will be randomized to one of the 2 arms. Patients belonging to study arm (Group II) will receive adjuvant radiotherapy 60 Gray, 30 fractions for 30 days over 6 weeks as routinely prescribed at Tata Memorial Center (TMC) and will receive the treatment within or by 6 weeks after surgery.

Both the groups (Group I and Group II) will be under regular follow-up with 3 monthly intervals for the first 2 years and 6 monthly for the next 3 years and once a year thereafter. At each follow-up, patients will be evaluated clinically for evidence of locoregional tumor recurrence. The locoregional recurrence-free survival will be calculated based on the difference between the date of randomization and the date of biopsy-proven recurrence. We will also record the overall survival in both groups. The quality of life will be assessed at each follow-up regular intervals using the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ H&N-35 ) and EORTC QLQ-C 30. The radiation toxicity will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) v4.0.

ELIGIBILITY:
Inclusion Criteria:

1. Post-operative early stage squamous cell carcinoma of the oral cavity (Oral Tongue, Buccal Mucosa, Floor of mouth). (pT1, pT2, N0 as defined in the AJCC Classification 8th edition.
2. Adequate surgery (Defined as wide local excision of the primary tumor with tumor-free margin ≥ 5mm and ipsilateral selective neck dissection addressing levels I-III at minimum.)
3. Written informed consent.
4. Age ≥18 years
5. Eastern Co-operative Oncology Group (ECOG) Performance Status 0-2
6. The depth of invasion (DOI) ≥ 5 mm.
7. Compliance to therapy and follow-up
8. The interval from surgery to adjuvant radiotherapy ≤ 6 weeks

Exclusion Criteria:

1. pT3/pT4 (as specified in the AJCC 8th edition).
2. Depth of invasion < 5mm.
3. Any neck nodal metastasis with or without extra nodal extension
4. Tumor-free margin < 5 mm
5. Non-squamous histology
6. Pregnant woman
7. Prior h/o any other malignancy in the last five years
8. Prior therapeutic irradiation of the head and neck.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
loco-regional recurrence free survival | Date of randomization to loco regional recurrence (date of proven biopsy date) or at the end of 36 months after recruitment of the last participant.
  Measures the number of local or regional recurrences in both arm over a defined time frame.

SECONDARY OUTCOMES:
Disease free survival | Calculated as difference of date of randomization to date of first documented recurrence or relapse, second primary or death or at the end of 36 months after recruitment of the last participant.
  time from the beginning of an intervention until patient experiences a recurrence, a new primary cancer or death.
Overall survival | Date of randomization to death from any cause or at the end of 36 months after recruitment of the last participant.
  Date of Randomization to death from any cause

OTHER OUTCOMES:
Quality of life Measurement | at Randomization, 3 months after completion of all treatments, 1 year, 2 years and 3 years after completion of all treatments.
  Measured using EORTC QLQ H&N-35 and EORTC QLQ-C 30
Acute and long-term Radiation toxicity rate | From the date of randomization until the date of first documented disease recurrence or date of death from any cause, assessed up to 36 months.
  The Common Terminology Criteria for Adverse Events (CTCAE V 4.0) will be used for assessing the Adverse events. The Radiation Therapy Oncology Group (RTOG) acute and late radiation morbidity scoring criteria will be used for assessing the radiotherapy related toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Sudhir V Nair, MS, MCh, Principal Investigator — Associate Professor
Locations (8):
- India (8):
  - Dr. B Barooah Cancer Institute, Guwahati, Assam
  - HCG Hospital, Ahmedabad, Gujarat
  - Kailash Cancer Hospital and Research Centre, Goraj, Gujarat
  - Sree Sankara Cancer Hospital, Bangalore, Karnataka
  - Mazumdar Shaw Medical Centre, Bangalore, Karnataka
  - Malabar Cancer Centre, Kannur, Kerala
  - Amrita Institute of Medical Sciences, Kochi, Kerala
  - Tata Memorial Centre, Mumbai, Maharashtra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thiagarajan S, Nair S, Nair D, Chaturvedi P, Kane SV, Agarwal JP, D'Cruz AK. Predictors of prognosis for squamous cell carcinoma of oral tongue. J Surg Oncol. 2014 Jun;109(7):639-44. doi: 10.1002/jso.23583. Epub 2014 Mar 12. PMID 24619660
- [Background] Dequanter D, Saint-Aubin N, Paesmans M, Badr-El-Din A, Lothaire P, Andry G. [Prognostic factors in epidermoid carcinoma of the mobile tongue classified as T1-T2]. Ann Otolaryngol Chir Cervicofac. 2001 Oct;118(5):315-22. French. PMID 11845040
- [Background] Kokemueller H, Rana M, Rublack J, Eckardt A, Tavassol F, Schumann P, Lindhorst D, Ruecker M, Gellrich NC. The Hannover experience: surgical treatment of tongue cancer--a clinical retrospective evaluation over a 30 years period. Head Neck Oncol. 2011 May 21;3:27. doi: 10.1186/1758-3284-3-27. PMID 21600000
- [Background] Ganly I, Patel S, Shah J. Early stage squamous cell cancer of the oral tongue--clinicopathologic features affecting outcome. Cancer. 2012 Jan 1;118(1):101-11. doi: 10.1002/cncr.26229. Epub 2011 Jun 29. PMID 21717431
- [Background] Gonzalez-Moles MA, Esteban F, Rodriguez-Archilla A, Ruiz-Avila I, Gonzalez-Moles S. Importance of tumour thickness measurement in prognosis of tongue cancer. Oral Oncol. 2002 Jun;38(4):394-7. doi: 10.1016/s1368-8375(01)00081-1. PMID 12076706
- [Background] Huang SF, Kang CJ, Lin CY, Fan KH, Yen TC, Wang HM, Chen IH, Liao CT, Cheng AJ, Chang JT. Neck treatment of patients with early stage oral tongue cancer: comparison between observation, supraomohyoid dissection, and extended dissection. Cancer. 2008 Mar 1;112(5):1066-75. doi: 10.1002/cncr.23278. PMID 18246535
- [Background] Shim SJ, Cha J, Koom WS, Kim GE, Lee CG, Choi EC, Keum KC. Clinical outcomes for T1-2N0-1 oral tongue cancer patients underwent surgery with and without postoperative radiotherapy. Radiat Oncol. 2010 May 27;5:43. doi: 10.1186/1748-717X-5-43. PMID 20504371
- [Background] Caramello P, Giacobbi D, Savoia D. [Identification of Pneumocystis carinii in a patient dying of AIDS]. G Batteriol Virol Immunol. 1985 Jul-Dec;78(7-12):171-7. Italian. PMID 3879892
- See also: SEER Cancer statistics review 1975-2010. National cancer institute — https://seer.cancer.gov/archive/csr/1975_2010/